CLINICAL TRIAL: NCT05485922
Title: A Randomized, Open-labelled, Crossover Study Confirming Performance of a Single-use Intermittent Micro-hole Zone Catheter in a Population of Adult Male Intermittent Catheter Users
Brief Title: Performance of a Single-use Intermittent Micro-hole Zone Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CP353
Record Dates: First submitted 2022-07-01; First posted 2022-08-03 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Urinary Incontinence; Retention, Urinary
MeSH Terms: conditions — Urinary Incontinence; Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Investigational device - intermittent catheter with a micro-hole zone (Experimental): A ready-to-use, sterile, hydrophilic-coated male catheter for intermittent catheterisation with a flexible tip and a micro-hole zone for urinary drainage in sizes CH12 and CH14. The catheterization was performed by a trained nurse.
  Interventions: Device: Investigational device - intermittent catheter with a micro-hole zone
- Comparator device - VaPro intermittent catheter (Active Comparator): Hollister VaPro, a single-use hydrophilic sleeved soft/flexible catheters in the sizes CH12 or CH14. The catheterization was performed by a trained nurse.
  Interventions: Device: Comparator device -VaPro intermittent catheter

INTERVENTIONS:
Device: Investigational device - intermittent catheter with a micro-hole zone — The investigational device was a urinary catheter for bladder drainage through the urethra. The product is for intermittent use.
  Arms: Investigational device - intermittent catheter with a micro-hole zone
Device: Comparator device -VaPro intermittent catheter — The comparator device is a urinary catheter for bladder drainage through the urethra. The product is for intermittent use.
  Arms: Comparator device - VaPro intermittent catheter

SUMMARY:
The goal of this randomized, controlled crossover study was to assess the performance of a new micro-hole zone catheter compared to a conventional 2-eyelet catheter in 42 male intermittent catheter users.

The main objective of this study was to demonstrate superiority of the micro-hole zone catheter in terms of number of flow-stop episodes and residual volume at first flow-stop, with the catheterization performed by a health care professional in a hospital setting compared to a conventional two-eyelet catheter.

DETAILED DESCRIPTION:
The investigation was a single-centre, randomized, controlled crossover study including 42 male participants comparing the performance of two intermittent catheters (IC).

The study included an information visit (visit 0) and two test visits (visit 1 and 2) in which one catheterization with either the investigational device or the comparator device, according to a randomization scheme, was performed by a health care professional in a hospital setting assessing flow stop episodes, bladder emptying and hematuria. There were 4-14 days between each test visit (visit 1 and 2) and visit 0 and 1 could be held on the same day.

ELIGIBILITY:
Inclusion Criteria:

1. Is Male
2. Is at least 18 years of age and has full legal capacity
3. Has given written informed consent
4. Has signed letter of authority (only DK)
5. Has used clean intermittent catheterisation CH12 or CH14 for at least one month
6. Use intermittent catheterisation as the primary bladder emptying method
7. Is able (assessed by investigator) and willing to follow study procedures

Exclusion Criteria:

1. Is participating in any other clinical study during this investigation
2. Has previous participated in this study
3. Has symptoms of urinary tract infection as judged by the investigator 4 Is an individual with history, suspected or showing signs of producing urine with excessive amount of mucus or large/clustered sediments or debris

5. Has any known allergies towards ingredients in the investigational device

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The device is a male catheter
Enrollment: 42 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cecilie Rovsing, MD, Principal Investigator — Sanos
Locations (1):
- Sanos Clinic, Gandrup, Denmark

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between August 2022 and November 2022, 42 users were recruited for the study from one site (Denmark) and encompassed the safety population.
Pre-assignment Details: The 42 recruited participants were randomized into the two intervention arms (the Intention to Treat, ITT), using a randomization sequence of 8. No participants were excluded or discontinued.
  All but one subject completed all visits due to data missing for one subject at visit 2. Accordingly, 41 catheterisation profiles were recorded for the investigational device and 42 for the comparator. No adverse events were reported.
Groups:
- Investigational Then Comparator: Participants were randomly assigned to the sequence of two intervention arms, in block sizes of 8.
  At the first intervention, one catheterization was performed with the investigational device, followed by a washout period of 4-14 days.
  At the second intervention, one catheterization was performed with the comparator device.
- Comparator Then Investigational: Participants were randomly assigned to the sequence of two intervention arms, in block sizes of 8.
  At the first intervention, one catheterization was performed with the comparator device, followed by a washout period of 4-14 days.
  At the second intervention, one catheterization was performed with the investigational device.
Period: Visit 1
Arm/Group | Investigational Then Comparator | Comparator Then Investigational
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0
Period: Visit 2
Arm/Group | Investigational Then Comparator | Comparator Then Investigational
Started | 21 | 21
Intention to Treat | 21 | 21
Completed | 21 (Data was missing for one participant at visit two in the investigational device group, but participant still completed the study.) | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total ITT Population Baseline Measures: Each investigation arm consisted of two test visits with 4-14 days of washout between each cross-over. On each visit, the participants underwent one intermittent catheterization performed by a trained nurse, through the urethra, draining the bladder, and testing a different intermittent catheter at each visit according to the randomization scheme.
  One catheterization with the investigational device which was a ready-to-use, sterile, hydrophilic-coated male catheter for intermittent catheterisation with a flexible tip and a micro-hole zone for urinary drainage in sizes CH12 and CH14. And one catheterization was with the comparator device which was a ready-to-use, sterile, hydrophilic-coated male catheter for intermittent catheterisation with a Hollister VaPro, in the sizes CH12 or CH14.
Arm/Group | Total ITT Population Baseline Measures
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 28
Age, Continuous [Mean (Full Range); unit: years] | 68 [41 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 42
Number of participants with neurogenic bladder dysfunction [Count of Participants; unit: Participants] | 13
Number of participants with non-neurogenic bladder dysfunction [Count of Participants; unit: Participants] | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Flow-stop Episodes
Description: Flow-stops were measured with a pressure sensor, which is an electronic device used for monitoring the hydrostatic pressure at the outlet of an intermittent urinary catheter during emptying.
  From a sensor curve, flow-stops were identified by two individually trained evaluators as a hydrostatic pressure peak coinciding with a urine flow-stop/ urine dripping (flowrate lower than 0,8 ml/sec).
  Results from both evaluators were compared and in case of discrepancy a discussion was performed to extenuate discrepancies and agree on a final interpretation of the curves.
Time Frame: Immediately after the procedure/catheterization
Population: The full analysis set
Measure: Mean (95% Confidence Interval); unit: Flow stop episodes
Groups:
- Investigational Device - Intermittent Catheter With a Micro-hole Zone (MHZ): A ready-to-use, sterile, hydrophilic-coated male catheter for intermittent catheterisation with a flexible tip and a micro-hole zone for urinary drainage. The external diameter is measured in millimeters (Charrière scale: Ch, CH) which were available in sizes CH12 and CH14. The catheterization was performed by a trained nurse.
  Investigational device - intermittent catheter with a micro-hole zone: The investigational device was a urinary catheter for bladder drainage through the urethra. The product is for intermittent use.
- Comparator Device - VaPro Intermittent Catheter: Hollister VaPro, a single-use hydrophilic sleeved soft/flexible catheters in the sizes CH12 or CH14 (which correspond to the external diameter measured in millimeters (Charrière scale: Ch, CH)). The catheterization was performed by a trained nurse.
  Comparator device -VaPro intermittent catheter: The comparator device is a urinary catheter for bladder drainage through the urethra. The product is for intermittent use.
Arm/Group | Investigational Device - Intermittent Catheter With a Micro-hole Zone (MHZ) | Comparator Device - VaPro Intermittent Catheter
Number analyzed (Participants) | 41 | 42
Flow stop episodes | 0.17 [0.06 to 0.45] | 1.09 [0.75 to 1.6]
Statistical Analysis 1: Comparison: Investigational Device - Intermittent Catheter With a Micro-hole Zone (MHZ) vs Comparator Device - VaPro Intermittent Catheter; Test type: Superiority — Number of flow-stop episodes will be analysed, in a generalized linier mixed model, with subject included as a random component. Evidence of superior effect will be concluded, if the lower 95% confidence limit of the risk ratio between comparator and investigational device, is more than 1; p < 0.05, Mixed Models Analysis; Risk Ratio (RR) = 0.16, 95% CI 2-sided [0.05 to 0.44]

2. Primary Outcome: Residual Urine at 1st Flow-stop
Description: The residual urine at 1st flow-stop during catheterization (performed by a nurse) represents the volume of urine left in the bladder, the first time the urine stops running out of the catheter during bladder emptying.
  Hence, the residual volume at 1st flow-stop was calculated as the total volume post catheterisation minus the volume at 1st flow-stop, derived from a catheterisation profile which was connected to a time-logged weighing [g].
Time Frame: When the first flow-stop appeared, the amount of voided urine was measured.
Population: The intention to treat population (full analysis set) constituted all randomized subjects with valid informed consent who was exposed to at least one product, and with valid information on at least one product with respect to the endpoints.
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Investigational Device - Intermittent Catheter With a Micro-hole Zone | Comparator Device - VaPro Intermittent Catheter
Number analyzed (Participants) | 42 | 42
mL | 5.10 [2.79 to 7.42] | 39.40 [19.92 to 58.89]
Statistical Analysis 1: Comparison: Investigational Device - Intermittent Catheter With a Micro-hole Zone vs Comparator Device - VaPro Intermittent Catheter; This was a superiority investigation in which the null hypothesis of the primary endpoints was to be rejected, at a 5% significance (alpha 0.05), to demonstrate the superiority of the investigational device; Test type: Superiority; p = 0.05, Mixed Models Analysis — The pass criteria were based on results analysing the 2 primary endpoints in a hierarchical fashion: rejecting the H0 on the first endpoint (Residual urine at first flow-stop) before continuing to the second (Number of flow-stop episodes); Mean Difference (Final Values) = 34.30, 95% CI 2-sided [14.69 to 53.91]

3. Primary Outcome: Number of Flow-stop Episodes
Description: Flow-stop episodes were determined as instances where the flow rate decreased to less than 0.8 mL/s for a period of at least two seconds. All episodes were detected by automatic thresholding, followed by manual inspection, where the intra-catheter pressure readings were used to support the assessment of a flow stop.
Time Frame: Immediately after catheterisation
Population: The intention to treat population (full analysis set) constituted all randomized subjects with a valid informed consent who was exposed to at least one product, and with valid information on at least one product with respect to the endpoints.
Measure: Number (95% Confidence Interval); unit: Flow stop episodes
Groups:
- Investigational Device: Participants were randomly assigned to the sequence of two intervention arms, in block sizes of 8.
  At the first intervention, one catheterization was performed with the investigational device, followed by a washout period of 4-14 days.
  At the second intervention, one catheterization was performed with the comparator device.
- Comparator Device: Participants were randomly assigned to the sequence of two intervention arms, in block sizes of 8.
  At the first intervention, one catheterization was performed with the comparator device, followed by a washout period of 4-14 days.
  At the second intervention, one catheterization was performed with the investigational device.
Arm/Group | Investigational Device | Comparator Device
Number analyzed (Participants) | 42 | 42
Flow stop episodes | 0.17 [0.06 to 0.45] | 1.09 [0.75 to 1.60]
Statistical Analysis 1: Comparison: Investigational Device vs Comparator Device; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — The pass criteria were based on the results analysing the two primary endpoints in a hierarchical fashion: rejecting the null hypothesis on the first endpoint (Residual urine at first flow-stop) before continuing to the second (Number of flow-stop episodes); p = 0.05, Mixed Models Analysis; Risk Ratio (RR) = 0.16, 95% CI 2-sided [0.05 to 0.44]

4. Other Pre Specified Outcome: Pressure Measurement at 1st Flow-stop Derived From a Catheterisation Profile.
Description: The intra-catheter pressure at the drainage holes, measured at 1st flow stop, was identified from a sensor curve.
Time Frame: When the first flow-stop appeared, the pressure at the drainage holes was measured
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: mbar
Arm/Group | Investigational Device | Comparator Device
Number analyzed (Participants) | 42 | 42
mbar | -16.14 [-22.50 to -9.79] | -111.83 [-153.4 to -70.26]
Statistical Analysis 1: Comparison: Investigational Device vs Comparator Device; The intra-catheter pressure at flow stop was analysed in a general linear mixed model with subject included as a random component; Test type: Superiority; p = 0.05, Mixed Models Analysis; Mean Difference (Final Values) = -95.69, 95% CI 2-sided [-137.69 to -53.70]

5. Other Pre Specified Outcome: Post-catheterisation Volume
Description: Post-catheterisation volume measured with a bladder Scanner assessed by the average of 3 consecutive measurements [mL]
Time Frame: Immediately after catheterisation
Population: as for outcome 3
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | Investigational Device | Comparator Device
Number analyzed (Participants) | 42 | 42
mL | 5.92 [-2.17 to 14.01] | 7.13 [-2.39 to 16.64]
Statistical Analysis 1: Comparison: Investigational Device vs Comparator Device; Test type: Other; p = 0.05, Mixed Models Analysis; Mean Difference (Final Values) = 1.21, 95% CI 2-sided [-11.10 to 13.51]

6. Post Hoc Outcome: Probability of a Positive Test for Hematuria
Description: Haematuria measured with a dipstick in the catheterised urine
Time Frame: Immediately after catheterisation
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: probability of positive test
Arm/Group | Investigational Device | Comparator Device
Number analyzed (Participants) | 42 | 42
probability of positive test | 0.10 [0.03 to 0.24] | 0.29 [0.17 to 0.45]
Statistical Analysis 1: Comparison: Investigational Device vs Comparator Device; Analyzed using a generalized linear mixed model, modelling the probability of a positive outcome. Evidence of effect in favour of the MHZC was concluded if the upper 95% confidence limit (CL) of the odds ratio, O.R. was less than 1; Test type: Superiority; p = 0.05, Mixed Models Analysis; Odds Ratio (OR) = 0.26, 95% CI 2-sided [0.07 to 0.96]

ADVERSE EVENTS:
Time Frame: Each participant was enrolled for 2x 1-14 days, thus a maximum of 28 days
Description: The relationship to the investigational or comparator products was collected. The safety population constituted the subjects who had given informed consent and were thus 42 participants.
  An adverse event was reported as either: "Not related", "Unlikely related", "Possibly related", "Probably related", or "Definitely related", to the comparator or to the investigational device.
Arm/Group | Investigational Device | Comparator Device
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/22/NCT05485922/Prot_SAP_000.pdf